CLINICAL TRIAL: NCT05881863
Title: To Investigate Airway Oxygen Concentrations During Rigid Bronchoscopy Procedures Performed With High Frequency Jet Ventilation
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: ANES-2022-31377
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Central Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
Thermal ablation (use of treatment modalities that generate heat) has become a widely used tool for treatment of central airway obstruction (e.g. laser, electrocautery, radiofrequency, and argon plasma coagulation). However, this method carries with it an increased risk for airway fire - a surgical fire that occurs in a patient's airway and could also include a fire in the attached breathing circuit. To decrease the risk of airway fire during mechanical ventilation with an endotracheal tube, the concentration of inspired oxygen (FiO2) is set below 40% while waiting for end tidal oxygen concentration (EtO2) to fall below 40% prior to starting thermal ablation. There is no published literature describing O2 concentration within the airways (AiO2) during jet ventilation with rigid bronchoscopy. The co-investigators of this study have recently collected data on AiO2 during rigid bronchoscopy using manual low frequency jet ventilation/high frequency jet ventilation with a period of apnea. The intent of this study is to measure the time taken for the central airway oxygen concentration to drop from 90 to 40% when the "laser mode" is activated on the Monsoon jet ventilator. Ventilation is continued during "laser mode."

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing rigid bronchoscopy for treatment of central airway obstruction at FV UMMC will be identified.
* 18 years or older
* Need rigid bronchoscopy as pre-determined by the interventional pulmonologist

Exclusion Criteria:

* Refusal to sign consent
* Pregnant patients
* Hemodynamic instability defined as continuous infusion of medication in order to support blood pressure and/or heart rate/rhythm
* Respiratory instability defined as SpO2<90% with >90% supplemental oxygen.
* Ineligible for rigid bronchoscopic intubation
* Latex allergy
* Evidence of fistulous airway
* Active Bronchopleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing rigid bronchoscopy for treatment of central airway obstruction at FV UMMC will be identified.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in seconds to AiO2 from 90 to 40% | baseline
  Time in seconds to AiO2 from 90 to 40% after activating laser mode on the monsoon jet ventilator.

SECONDARY OUTCOMES:
Differences in time to laser mode AiO2 | baseline
  Differences in time to laser mode AiO2 between trachea and left and right mainstem bronchi.

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Setty, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States